CLINICAL TRIAL: NCT02613806
Title: Effects of Dexmedetomidine on Cough Response and Postoperative Recovery Quality in Patients Undergoing Thyroid Surgery With General anesthesia---a Randomized Control Double-Blind Clinical Trial
Brief Title: Effects of Dexmedetomidine on Cough Response and Postoperative Recovery Quality in Patients Undergoing Thyroid Surgery With General Anesthesia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Min Su, The Department of Anesthesia and Pain Medicine, First Affiliated Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CYYYMZK-08
Record Dates: First submitted 2015-11-23; First posted 2015-11-25 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-11

CONDITIONS: Coughing Response; Thyroid Surgery; General Anesthesia
Keywords: Dexmedetomidine; Coughing Response; Postoperative Recovery Quality; Thyroid Surgery
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- D group (dexmedetomidine) (Experimental): Dexmeditomidine 0.2 ug/kg·h will be administered to participants by intravenous infusion with microperfusion pump at the beginning of the surgery,and continued till end of surgery.
  Interventions: Drug: Dexmeditomidine
- C group (saline) (Active Comparator): The patients received equal volume normal saline by intravenous infusion at the beginning of the surgery,and continued till end of surgery.
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Dexmeditomidine — Dexmeditomidine 0.2 ug/kg·h will be administered to participants by intravenous infusion at the beginning of the surgery,and continued till end of surgery.
  Arms: D group (dexmedetomidine)
Drug: normal saline — Isovolumetric normal saline will be administered to participants by intravenous infusion at the beginning of the surgery,and continued till end of surgery.
  Arms: C group (saline)

SUMMARY:
Coughing is a common adverse reaction of thyroid surgery,which could result in postoperative bleeding.Postoperative bleeding is a serious and potentially life-threatening complication，which could result in acute upper airway obstruction due to neck hematoma and increase the need for re-operation.The purpose of this study is to investigate whether dexmedetomidine can reduce the incidence of postoperative coughing and contribute to postoperative recovery in patients undergoing tyroid surgery with general anesthesia.

DETAILED DESCRIPTION:
Thyroid surgery is a common clinical surgery,the incidence of postoperative coughing is up to 32.4%.Coughing response could result in postoperative bleeding,even cause respiratory tract obstruction,affect patients' postoperative recovery .Dexmedetomidine,an α2 adrenergic agonist,has hypnotic,analgesic, anxiolytic,antisympathetic effects,which could facilitate the sedation of patients while maintaining their consciousness and keep respiration and circulation stable .For these benefits,dexmedetomidine was widely used for general anesthesia.However,whether dexmedetomidine can reduce the incidence of postoperative coughing is unclear.Therefore,the investigators conduct this randomized controlled double-blind trial,to investigate the effects of dexmedetomidine on coughing and postoperative recovery quality in patients undergoing tyroid surgery with general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

1. Aged from 18 to 65 years old
2. American Society of Anesthesiologists (ASA) physical statusⅠor Ⅱ
3. Diagnosed by B ultrasonic or tissue biopsy show that patients thyrophyma,thyroid cancer,thyroid nodule,etc,who need to accept thyroid surgery

Exclusion Criteria:

1. large goiter or hyperthyroidism
2. Preoperative coughing caused by primary diseases of patients
3. Ⅱdegrees above atrioventricular block
4. Allergy to anesthesia
5. History of diabetes
6. Pregnant women
7. Serious mental disease
8. History of alcohol or drug abuse
9. Severe heart renal or liver dysfunction
10. The presence of an upper respiratory infection
11. Asthma
12. Anticipated difficult airway

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 118 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
the incidence of coughing | within 48 hours postoperatively
  coughing will be observed

SECONDARY OUTCOMES:
coughing on a four-point scale | within 48 hours postoperatively
  coughing on a four-point scale will be measured within 48 hours postoperatively
the eyes opening time | within 48 hours postoperatively
  the eyes opening time will be observed
the time of extubation | within 48 hours postoperatively
  the time of extubation will be recorded
visual analogue scale (VAS) | at 30 minutes after extubation
  visual analogue scale will be measured at 30 minutes after extubation
sedation-agitation scale(SAS) | at 30 minutes after extubation
  sedation-agitation scale will be measured at 30 minutes after extubation

CONTACTS AND LOCATIONS:
Overall Officials: Su Min, Principal Investigator — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- The First Affliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Background] Bergese SD, Khabiri B, Roberts WD, Howie MB, McSweeney TD, Gerhardt MA. Dexmedetomidine for conscious sedation in difficult awake fiberoptic intubation cases. J Clin Anesth. 2007 Mar;19(2):141-4. doi: 10.1016/j.jclinane.2006.07.005. PMID 17379129
- [Background] Kaya FN, Yavascaoglu B, Turker G, Yildirim A, Gurbet A, Mogol EB, Ozcan B. Intravenous dexmedetomidine, but not midazolam, prolongs bupivacaine spinal anesthesia. Can J Anaesth. 2010 Jan;57(1):39-45. doi: 10.1007/s12630-009-9231-6. Epub 2009 Dec 29. PMID 20039221
- [Background] Kiray A, Naderi S, Ergur I, Korman E. Surgical anatomy of the internal branch of the superior laryngeal nerve. Eur Spine J. 2006 Sep;15(9):1320-5. doi: 10.1007/s00586-005-0006-7. Epub 2006 Jan 5. PMID 16402208
- [Background] Kamibayashi T, Maze M. Clinical uses of alpha2 -adrenergic agonists. Anesthesiology. 2000 Nov;93(5):1345-9. doi: 10.1097/00000542-200011000-00030. No abstract available. PMID 11046225
- [Background] Bekker A, Haile M, Kline R, Didehvar S, Babu R, Martiniuk F, Urban M. The effect of intraoperative infusion of dexmedetomidine on the quality of recovery after major spinal surgery. J Neurosurg Anesthesiol. 2013 Jan;25(1):16-24. doi: 10.1097/ANA.0b013e31826318af. PMID 22824921
- [Background] Ham SY, Kim JE, Park C, Shin MJ, Shim YH. Dexmedetomidine does not reduce emergence agitation in adults following orthognathic surgery. Acta Anaesthesiol Scand. 2014 Sep;58(8):955-60. doi: 10.1111/aas.12379. PMID 25132201